CLINICAL TRIAL: NCT01913496
Title: Development of Internet Web Application and Evaluation of Its Impact as a Tool in Promoting Healthy Lifestyle Indicators in Adults
Brief Title: Development of Web Application and Evaluation Its Impact on Healthy Lifestyle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew University of Jerusalem (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Jenny Naimark, PhD student, Hebrew University of Jerusalem
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: eBalance
Record Dates: First submitted 2013-07-25; First posted 2013-08-01 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Lifestyle
Keywords: web application; nutrition knowledge; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (Placebo Comparator): standard care ,without the web application ebalance
  Interventions: Other: ebalance
- ebalance (Active Comparator): using the ebalance application for 14 weeks
  Interventions: Other: ebalance

INTERVENTIONS:
Other: ebalance — using the ebalance application for 14 weeks

SUMMARY:
The study is planned for people who would like to reduce or maintain their weight and keep a healthy life style .After signing an informed consent, participants will be divided randomly into two groups :control group and an intervention group that will get the application (eBalance ). Participants will be followed for 12 weeks.

DETAILED DESCRIPTION:
Primary objective: to develop a web application based on energy balance and evaluates its effectiveness in promoting healthy lifestyle habits versus a control group.

Secondary objectives:

1. To evaluate the frequency and convenient of usage of the internet intervention
2. To test the impact of the intervention on nutrition knowledge, diet quality and physical activity
3. To evaluate the effect of the intervention on weight management status

ELIGIBILITY:
Inclusion Criteria:

* People aged more than 18 years
* Web and e-mail experience
* Interested in either reducing weight or maintaining a healthy lifestyle

Exclusion Criteria:

* without any mail experience
* pregnancy
* involvement in other diet programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
weight | 14 weeks
  measuring weight at baseline and end of 14 weeks

SECONDARY OUTCOMES:
duration of physical activity | 14 weeks
  at baseline and end of study
Nutrition knowledge | 14 weeks
  questionnaire at baseline and end of study
waist circumference | 14 weeks
  waist circumference will be measured at baseline and end of 14 weeks
height | 14 weeks
  height will be measured at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Naimark, PhD student, Principal Investigator — Hebrew University
Locations (1):
- Hebrew University, Jerusalem, Israel

REFERENCES:
- [Derived] Safran Naimark J, Madar Z, Shahar DR. The impact of a Web-based app (eBalance) in promoting healthy lifestyles: randomized controlled trial. J Med Internet Res. 2015 Mar 2;17(3):e56. doi: 10.2196/jmir.3682. PMID 25732936